CLINICAL TRIAL: NCT05239182
Title: A Phase 2 Study of 9-ING-41, a Glycogen Synthase Kinase 3-beta (GSK-3β) Inhibitor, Combined With Retifanlimab, a PD-1 Inhibitor, Plus Gemcitabine/Nab-Paclitaxel as Frontline Therapy for Patients With Advanced Pancreatic Adenocarcinoma (RiLEY)
Brief Title: 9-ING-41 Plus Retifanlimab and Gemcitabine/Nab-Paclitaxel in Patients With Advanced Pancreatic Adenocarcinoma
Acronym: RiLEY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Backbone chemo regimen of gemzar/abraxane no longer most favorable treatment for pancreatic cancer patients.
Sponsor: Anwaar Saeed (Other)
Collaborators: Actuate Therapeutics Inc. (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Anwaar Saeed, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-194
Record Dates: First submitted 2022-01-26; First posted 2022-02-14 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: glycogen biosynthesis; Glycogen synthase kinase-3 (GSK-3); NF-κB pathway
MeSH Terms: interventions — 3-(5-fluorobenzofuran-3-yl)-4-(5-methyl-5H-(1,3)dioxolo(4,5-f)indol-7-yl)-pyrrole-2,5-dione; Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 9-ING-41 plus Retifanlimab plus Gem/Abraxane (Experimental): * intravenous (IV) infusion of nab-paclitaxel at a dose of 125 mg per square meter, followed by an infusion of gemcitabine according to the gemcitabine label at a dose of 1000 mg per square meter, on days 1, 8, 15 of a 28-day cycle.
  * Retifanlimab 500 mg IV on day 1 of a 28-day cycle. (Retifanlimab will be administered following gemcitabine/nab-paclitaxel.)
  * 9-ING-41 administered at a dose of 9.3 mg/kg by IV infusion twice weekly on Days 1 and 4 of each week of a 28-day cycle. (9-ING-41 will be administered following retifanlimab.)
  Interventions: Drug: 9-ING-41; Drug: Retifanlimab; Drug: Gemcitabine; Drug: Abraxane

INTERVENTIONS:
Drug: 9-ING-41 — 9-ING-41 is a small molecule potent selective GSK-3β inhibitor
Drug: Retifanlimab — Humanized, hinge-stabilized, IgG4κ monoclonal antibody that recognizes human PD-1.
  Other Names: INCMGA00012
Drug: Gemcitabine — cytotoxic chemotherapy agent
Drug: Abraxane — cytotoxic chemotherapy agent

SUMMARY:
This trial examines how Pancreatic Adenocarcinoma reacts to the addition of 9-ING-41 and retifanlimab to the standard of care chemotherapy treatment, to see if using this combination will help and is able to effect disease progression.

DETAILED DESCRIPTION:
Given the role of GSK-3β in immune regulation, the combination of GSK-3β inhibition with PD 1 inhibition may be expected to provide synergistic anti-tumor efficacy. The excellent safety profile of 9-ING-41, along with preclinical and clinical evidence of anti-tumor activity in pancreatic cancer, provides a strong rationale to evaluate the efficacy of 9-ING-41 in combination with a PD 1 inhibitor plus standard chemotherapy (gemcitabine/nab-paclitaxel) as frontline therapy for patients with advanced PDAC.

The combination of 9-ING-41 and retifanlimab with gemcitabine/nab-paclitaxel has not previously been administered to human subjects. In the 1801 study, 9-ING- 41 has been administered in combination with various chemotherapy regimens including gemcitabine/nab-paclitaxel, with one 9-ING-41-related SAE (transient visual change) documented to date. Retifanlimab alone has been well-tolerated when administered for up to 2 years in patients with anal cancer. Overall, based on previous nonclinical and clinical experience, both of these agents appear to have an acceptable safety profile and do not appear to have significant overlapping toxicities. However, it is possible that when they are administered together and in combination with gemcitabine/nab-paclitaxel, more frequent or severe AEs, or new AEs not previously observed with any of these agents administered alone, may occur.

It is not known if administration of 9-ING-41 and retifanlimab will act synergistically to provide increased anti-tumor activity compared to gemcitabine/nab-paclitaxel alone. Subjects in this study should not expect to benefit directly by their participation in the study. The data collected in this study may benefit future cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily written informed consent and willingness/ability to comply with the protocol requirements
* Has pathologically confirmed advanced, recurrent, or metastatic pancreatic cancer AND is previously untreated with systemic agents in the advanced/metastatic setting.
* Must have at least 1 measurable lesion per RECIST v1.1. Lesions that are radiated should not count as target lesions unless there is evidence of growth post radiation on a subsequent scan prior to trial enrollment.
* Must have available archived tumor tissue at study entry (metastatic tissue preferred to primary tissue)
* Adequate bone marrow function: absolute neutrophil count (ANC) ≥ 1000/mL; hemoglobin ≥ 8.5 g/dL, platelets ≥ 100,000/mL.
* Adequate liver function: transaminases (aspartate aminotransferase/ alanine aminotransferase, AST/ALT) and alkaline phosphatase ≤ 2.5 x ULN (≤ 5 X the upper limit of normal (ULN) in the setting of liver metastasis or infiltration with malignant cells); bilirubin ≤ 1.5 x ULN.
* Adequate renal function: creatinine clearance CrCl > 60 mL/min measured or calculated by Cockcroft- Gault (C-G) equation (estimated glomerular filtration rate [eGFR] can also be used in place of CrCl).
* Serum amylase and lipase ≤ 1.5 x ULN
* Eastern Co-operative Oncology Group (ECOG) performance status (PS) 0 - 1
* Has received the final dose of any of the following treatments/ procedures within the specified minimum intervals before first dose of study drug: Focal radiation therapy - 7 days Surgery with general anesthesia - 7 days Surgery with local anesthesia - 7 days

Exclusion Criteria:

* Is pregnant or lactating.
* Is known to be hypersensitive to any of the components or metabolites of 9-ING-41 or to the excipients used in its formulation, or known sensitivity to one of the chemotherapeutic agents or to the PD-1 inhibitor.
* History of receiving prior treatment with any anti-PD-1, PD-L1 or PD-L2 agent.
* Has endocrine or acinar pancreatic carcinoma.
* Has not recovered from clinically significant toxicities as a result of prior anticancer therapy, except alopecia, anemia not requiring transfusion support and infertility. Recovery is defined as ≤ Grade 1 or baseline severity per Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5.0).
* Has significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, or stroke within 6 months of the first dose of 9-ING-41, or cardiac arrhythmia requiring medical treatment detected at screening.
* Has had a myocardial infarction within 12 weeks of the first dose of 9-ING-41 or has electrocardiogram (ECG) abnormalities that are deemed medically relevant by the investigator or study medical coordinator.
* Has symptomatic rapidly progressive brain metastases or leptomeningeal involvement as assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI). Patients with stable brain metastases or leptomeningeal disease or slowly progressive disease are eligible provided that they have not required new treatments for this disease in a 28-day period before the first dose of study drug, and anticonvulsants and steroids are at a stable dose for a period of 14 days prior to the first dose of study drug.
* Has had major surgery (not including placement of central lines) within 7 days prior to study entry or is planned to have major surgery during the course of the study (major surgery may be defined as any invasive operative procedure in which an extensive resection is performed, e.g., a body cavity is entered, organs are removed, or normal anatomy is altered).
* Has any medical and/or social condition that, in the opinion of the investigator would preclude study participation.
* Has received an investigational anti-cancer drug in the 14-day period before the first dose of study drug (or within 5 half-lives if longer) or is currently participating in another interventional clinical trial.
* Has a current malignancy other than pancreatic cancer.
* Known immunodeficiency syndrome or active autoimmune disease or requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg/day of prednisone or equivalent).
* Evidence of interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis.
* Palliative radiation therapy administered within 1 week of first dose of study treatment or radiation therapy that is > 30 Gy within 6 months of the first dose of study treatment.
* Has received systemic antibiotics ≤ 7 days prior to the first dose of study drug.
* History of organ transplant, including allogeneic stem cell transplantation.
* Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures (eg, antihistamines and corticosteroids).
* Known allergy or hypersensitivity to any component of retifanlimab or formulation components.
* Has received a live vaccine within 28 days of the planned start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anwaar Saeed, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Kansas University Cancer Center, Fairway, Kansas
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw G, Cavalcante L, Giles FJ, Taylor A. Elraglusib (9-ING-41), a selective small-molecule inhibitor of glycogen synthase kinase-3 beta, reduces expression of immune checkpoint molecules PD-1, TIGIT and LAG-3 and enhances CD8+ T cell cytolytic killing of melanoma cells. J Hematol Oncol. 2022 Sep 14;15(1):134. doi: 10.1186/s13045-022-01352-x. PMID 36104795

RESULTS

PARTICIPANT FLOW:
Groups:
- 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane: * intravenous (IV) infusion of nab-paclitaxel at a dose of 125 mg per square meter, followed by an infusion of gemcitabine according to the gemcitabine label at a dose of 1000 mg per square meter, on days 1, 8, 15 of a 28-day cycle.
  * Retifanlimab 500 mg IV on day 1 of a 28-day cycle. (Retifanlimab will be administered following gemcitabine/nab-paclitaxel.)
  * 9-ING-41 administered at a dose of 9.3 mg/kg by IV infusion twice weekly on Days 1 and 4 of each week of a 28-day cycle. (9-ING-41 will be administered following retifanlimab.)
    9-ING-41: 9-ING-41 is a small molecule potent selective GSK-3β inhibitor
  Retifanlimab: Humanized, hinge-stabilized, IgG4κ monoclonal antibody that recognizes human PD-1.
  Gemcitabine: cytotoxic chemotherapy agent
  Abraxane: cytotoxic chemotherapy agent
Period: Overall Study
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.14286 (5.607939)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex is 'Unknown' for one patient.
  Participants
    number analyzed (Participants) | 6
    Female | 3
    Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: Percentage of patients with stable disease (SD), Complete Response (CR), or Partial Response (PR) for ≥16 weeks during treatment. Per RECIST v1.1, (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to approximately 11 months from baseline
Population: Treated patients who were radiologically evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 6
percentage of patients | 100

2. Secondary Outcome: Best Response
Description: Number of patients with Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) per RECIST v1.1 Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 12 months (from enrollment)
Population: Treated patients who were radiologically evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 6
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 4
  Progressive Disease | 0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Percentage of patients with Complete Response (CR) or Partial Response (PR) per RECIST v1.1 Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 12 months (from enrollment)
Population: Treated patients who were radiologically evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 6
percentage of patients | 33

4. Secondary Outcome: Adverse Events and Serious Adverse Events
Description: Number of participants with overall treatment-related adverse events (AE) and/or serious adverse events (SAE) at least possibly related as assessed by CTCAE v5.0.
Time Frame: Up to 12 months (from enrollment)
Population: All patients who receive at least one dose of 9-ING-41
Measure: Number; unit: participants
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 7
participants
  Alanine aminotransferase increased | 2
  Alopecia | 2
  Anemia | 5
  Anorexia | 1
  Aspartate aminotransferase increased | 1
  Ataxia | 1
  Blurred vision | 1
  Colitis | 1
  Constipation | 1
  Diarrhea | 5
  Dizziness | 1
  Edema limbs | 3
  Eye disorder | 1
  Fatigue | 4
  Febrile neutropenia | 1
  Fever | 2
  Flu like symptoms | 1
  Headache | 1
  Hyperkalemia | 1
  Hypokalemia | 2
  Hypomagnesemia | 2
  Hyponatremia | 1
  Mucositis oral | 3
  Nail changes | 1
  Nail discoloration | 1
  Nausea | 4
  Neutrophil count decreased | 4
  Papulopustular rash | 1
  Periorbital Dermatitis | 1
  Peripheral motor neuropathy | 1
  Peripheral sensory neuropathy | 1
  Platelet count decreased | 3
  Pruritus | 3
  Rash maculo-papular | 2
  Sepsis | 2
  Skin and subcutaneous tissue disorders - Other, specify | 1
  Syncope | 1
  Throat pain | 1
  Vomiting | 2
  Weight loss | 4
  White blood cell decreased | 2

5. Secondary Outcome: Duration of Response (DOR)
Description: Time from documentation of tumor response to disease progression. Per RECISIT v1.1, Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 12 months (from enrollment)
Population: Treated patients who were radiologically evaluable.
Measure: Median (Full Range); unit: months
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 2
months | 5.273 [4.862 to 5.684]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from study enrollment until objective tumor progression or death. Per RECISIT v1.1, Progressive Disease (PD) is ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 12 months (from enrollment)
Population: Treated patients evaluable for radiologic response.
Measure: Median (Full Range); unit: months
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 6
months | 6.785481 [4.970569 to 8.69]

7. Secondary Outcome: Overall Survival (OS)
Description: Time patients are alive from study enrollment to death from any cause.
Time Frame: Up to 24 months
Population: All study enrolled participants.
Measure: Median (Full Range); unit: months
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
Number analyzed (Participants) | 7
months | 10.72596 [6.965337 to 20.40549]

ADVERSE EVENTS:
Time Frame: Adverse Events data collected for up to 12 months. All-Cause Mortality data collected for up to 24 months
Arm/Group | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane
All-Cause Mortality (participants affected / at risk) | 4/7
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane (N=7)
Blood bilirubin increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Sepsis (Infections and infestations) | 2
Colitis (Gastrointestinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 9-ING-41 Plus Retifanlimab Plus Gem/Abraxane (N=7)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Ascites (Hepatobiliary disorders) | 1
Aspartate aminotransferace (Investigations) | 2
Ataxia (Nervous system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bilateral peripheral neuropathy (Nervous system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 5
Edema limbs (Vascular disorders) | 3
Fall (General disorders) | 1
Fatigue (General disorders) | 4
Febrile neutropenia (Investigations) | 1
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hyperkalemia (Investigations) | 1
Hypokalemia (Investigations) | 2
Hypomagnesemia (Investigations) | 2
Hyponatremia (Investigations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Neutrophil count decreased (Investigations) | 4
Non-cardiac chest pain (General disorders) | 1
Pain in extremity (General disorders) | 1
Pancreatic fistula (Gastrointestinal disorders) | 1
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Periorbital Dermatitis (Skin and subcutaneous tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1
Transient visual changes- things appearing darker (Eye disorders) | 2
Urine discoloration (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Weight loss (General disorders) | 4
White blood cell decreased (Investigations) | 2
Dizziness (Nervous system disorders) | 1
Dysgeusia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT05239182/Prot_SAP_000.pdf